CLINICAL TRIAL: NCT04719481
Title: The Reduction Effect of Oral Pravastatin on Acute Phase Response of Intravenous Zoledronic Acid: a Real-world Study
Brief Title: Pravastatin Reduces Acute Phase Response of Zoledronic Acid
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2020180
Record Dates: First submitted 2021-01-06; First posted 2021-01-22 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Postmenopausal Osteoporosis
Keywords: acute phase response; zoledronic acid; pravastatin
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Acute-Phase Reaction | interventions — Pravastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pravastatin 80mg/d (Experimental): Oral administration of pravastatin at 1 h before zoledronic acid infusion, 24 h and 48 h after zoledronic acid infusion
  Interventions: Drug: Pravastatin Sodium 80 MG
- placebo (Placebo Comparator): Oral administration of placebo at 1 h before zoledronic acid infusion, 24 h and 48 h after zoledronic acid infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pravastatin Sodium 80 MG — daily oral administration of 80mg
  Other Names: Meibailezhen
  Arms: pravastatin 80mg/d
Drug: Placebo — daily oral administration
  Other Names: Meibailezhen placebo
  Arms: placebo

SUMMARY:
Acute phase response (APR) is one of the most common adverse events in osteoporosis with zoledronic acid treatment. It's reported that this reaction is related to the blockade of the mevalonate pathway, leading to isopentenyl pyrophosphate (IPP) accumulation. And the latter can active γδT cells in the circulation, resulting in inflammatory cytokine release. Statins can inhibit the conversion of HMG-CoA to mevalonate that may reduce the accumulation of IPP. Therefore, it is possible that statins can be taken in advance to reduce APR caused by zoledronic acid infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese Han ethnic postmenopausal women.
2. Bone mineral density values of less than 2.5 standard deviations (SD) below the normal adult mean.
3. Willing to participate in this study.

Exclusion Criteria:

1. Prior treatment with biphosphonates (oral or intravenous).
2. Fever and/or any viral or bacterial infections within 30 days prior to randomization.
3. Patients with evidence of any cancer or with a history of cancer.
4. Contraindication to zoledronic acid:

   Known hypersensitivity to zoledronic acid or other bisphosphonate or zoledronic acid formulation (excipients); Serum calcium level < 2.13 mmol/L (8.5 mg/dL), free serum calcium level <0.95 mmol/L (3.8 mg/dL) or untreated hypocalcemia; Childbearing or child-breastfeeding women; Creatinine clearance < 35 mL/min;

   Restrictions:

   Patients currently receiving aminoglycoside, diuretics or thalidomide.
5. Contraindication to pravastatin:

   Known hypersensitivity to pravastatin or other excipients in pravastatin sodium formulation.

   Restrictions:

   Patients with severe liver insufficiency, history of severe liver insufficiency, active liver disease or continuously elevated transaminase; Patients with severe renal insufficiency or history of severe renal insufficiency; Patients currently receiving fibrates (e.g., bezafibrate), immunosuppressive drug (e.g., cyclosporine) or niacin.
6. Any physiological or medical condition which, in the opinion of the investigator, would preclude the participant from this trail.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute phase response | 0-72 hours
  Effect of oral pravastatin on the incidence of acute phase response within 72 hours after zoledronic acid infusion

SECONDARY OUTCOMES:
Occurrence time of fever | from 8:00 a.m. to 8:00 p.m. with interval of 4 hours in Day -2 and Day -1, from 9:00 a.m. to 9:00 p.m. with interval of 3 hours in Day 0, 1, 2, 3. It should be recorded when fever occurs in other time.
  Effect of oral pravastatin on the occurrence time of fever after zoledronic acid infusion
Severity of fever | from 8:00 a.m. to 8:00 p.m. with interval of 4 hours in Day -2 and Day -1, from 9:00 a.m. to 9:00 p.m. with interval of 3 hours in Day 0, 1, 2, 3. It should be recorded when fever occurs in other time.
  Effect of oral pravastatin on the severity of fever (body temperature) after zoledronic acid infusion.
Occurrence time of pain | from 8:00 a.m. to 8:00 p.m. with interval of 4 hours in Day -2 and Day -1, from 9:00 a.m. to 9:00 p.m. with interval of 3 hours in Day 0, 1, 2, 3. It should be recorded when pain occurs in other time.
  Effect of oral pravastatin on the occurrence time of pain after zoledronic acid infusion
Severity of pain | from 8:00 a.m. to 8:00 p.m. with interval of 4 hours in Day -2 and Day -1, from 9:00 a.m. to 9:00 p.m. with interval of 3 hours in Day 0, 1, 2, 3. It should be recorded when pain occurs in other time.
  Effect of oral pravastatin on the severity of pain (visual analogue scale, VAS) after zoledronic acid infusion
Frequency of acetaminophen usage after zoledronic acid infusion | within 72 hours after zoledronic acid infusion
  To compare the frequency of acetaminophen within 72 hours after zoledronic acid infusion between pravastatin arm and placebo arm.
Amount of acetaminophen usage after zoledronic acid infusion | within 72 hours after zoledronic acid infusion
  To compare the amount of acetaminophen within 72 hours after zoledronic acid infusion between pravastatin arm and placebo arm.
White blood cells | baseline and 48 hours after infusion
  To compare the changes in white blood cells (WBC) count within 48 hours after zoledronic acid infusion between pravastatin arm and placebo arm.
C reaction protein | baseline and 48 hours after infusion
  To compare the changes in C reaction protein (CRP) within 48 hours after zoledronic acid infusion between pravastatin arm and placebo arm.
interferon-γ expression | baseline and 48 hours after infusion
  To compare the changes in interferon-γ (IFN-γ) within 48 hours after zoledronic acid infusion between pravastatin arm and placebo arm.
interleukin-6 expression | baseline and 48 hours after infusion
  To compare the changes in interleukin-6 (IL-6) within 48 hours after zoledronic acid infusion between pravastatin arm and placebo arm.
γδT cells activation | baseline and 48 hours after infusion
  To compare the changes in count of γδT cells activation within 48 hours after zoledronic acid infusion pravastatin arm and placebo arm.
Adverse event occurrence | 0-10 days
  The occurrence of adverse event within 10 days after zoledronic acid infusion

CONTACTS AND LOCATIONS:
Overall Officials: Chunli Song, M.D.; Ph. D., Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sieber P, Lardelli P, Kraenzlin CA, Kraenzlin ME, Meier C. Intravenous bisphosphonates for postmenopausal osteoporosis: safety profiles of zoledronic acid and ibandronate in clinical practice. Clin Drug Investig. 2013 Feb;33(2):117-22. doi: 10.1007/s40261-012-0041-1. PMID 23184667
- [Background] Hewitt RE, Lissina A, Green AE, Slay ES, Price DA, Sewell AK. The bisphosphonate acute phase response: rapid and copious production of proinflammatory cytokines by peripheral blood gd T cells in response to aminobisphosphonates is inhibited by statins. Clin Exp Immunol. 2005 Jan;139(1):101-11. doi: 10.1111/j.1365-2249.2005.02665.x. PMID 15606619
- [Background] Sireci G, Espinosa E, Di Sano C, Dieli F, Fournie JJ, Salerno A. Differential activation of human gammadelta cells by nonpeptide phosphoantigens. Eur J Immunol. 2001 May;31(5):1628-35. doi: 10.1002/1521-4141(200105)31:53.0.CO;2-T. PMID 11465120
- [Background] Schneiders FL, Huijts CM, Reijm M, Bontkes HJ, Verheul HMW, de Gruijl TD, van der Vliet HJ. The effects of systemic treatment with aminobisphosphonates and statins on circulating Vgamma9Vdelta2-T cells in patients with advanced cancer. Immunobiology. 2018 Feb;223(2):171-177. doi: 10.1016/j.imbio.2017.10.029. Epub 2017 Oct 16. PMID 29055564
- [Derived] Liu Q, Han G, Li R, Fan D, Du G, Zhang M, Tao L, Li H, Liu D, Song C. Reduction effect of oral pravastatin on the acute phase response to intravenous zoledronic acid: protocol for a real-world prospective, placebo-controlled trial. BMJ Open. 2022 Jul 13;12(7):e060703. doi: 10.1136/bmjopen-2021-060703. PMID 35831045